CLINICAL TRIAL: NCT06035835
Title: Probiotics and Breastmilk Are Associated With a Decreased Risk of Atopic Dermatitis in Very Low Birth Weight Premature Infants
Brief Title: Probiotics and Breastmilk Decrease Risk of Atopic Dermatitis in Premature Infants
Status: Completed | Type: Observational
Sponsor: José Uberos Fernández (Other)
Responsible Party: Sponsor-Investigator, José Uberos Fernández, Head of Unit Care Neonatology, Principal Investigator, Clinical Professor, Hospital Clinico Universitario San Cecilio
Organization: Hospital Clinico Universitario San Cecilio (Other)
Other Study IDs: BM-2022-12-0144.R2
Record Dates: First submitted 2023-07-26; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis
Keywords: Probiotics; Human breastmilk; newborn; very low birth weight; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Lacteol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Probiotic 1: Administration Lacticaseibacillus rhamnosus (L. Rhamnosus) ATCC 53103 (109 UFC/day) in very low birth weight since start at the first enteral feed until 35 week Postmenstrual age
  Interventions: Combination Product: Lacticaseibacillus rhamnosus
- Probiotic 2: Administration Lactobacillus acidophilus (L. acidophilus) ATCC 4356 (109 UFC/12 h)+Bifidobacterium bifidum (B. bifidum) ATCC 15696 (109 UFC/12 h) in very low birth weight since start at the first enteral feed until 35 week Postmenstrual age
  Interventions: Combination Product: Lactobacillus acidophilus + Bifidobacterium bifidum
- No probiotic: No suplementation diet with probiotic

INTERVENTIONS:
Combination Product: Lacticaseibacillus rhamnosus — Administration Lacticaseibacillus rhamnosus (L. Rhamnosus) ATCC 53103 (109 UFC/day)
  Groups: Probiotic 1
Combination Product: Lactobacillus acidophilus + Bifidobacterium bifidum — Administration Lactobacillus acidophilus (L. acidophilus) ATCC 4356 (109 UFC/12 h)+Bifidobacterium bifidum (B. bifidum) ATCC 15696 (109 UFC/12 h)
  Groups: Probiotic 2

SUMMARY:
The purpose of this study is assess if the use of probiotic in very low weight could be other benefits a long time, as reduce atopic disease in this children.

DETAILED DESCRIPTION:
In this study, the investigators analyse the influence of nutrition during the early neonatal period on the development and prevention of atopic dermatitis (AD) in children with a history of very low birth weight (VLBW). A retrospective cohort study was performed of VLBW preterm infants to assess the risk of their developing AD during childhood, according to nutrition with breastmilk and/or probiotic supplementation during the neonatal period. The analysis focused on nutritional and early childhood follow-up data for 437 newborns, of whom 184 received probiotics up to 36 weeks postmenstrual age.

The neonatal history of the patients was consulted in their electronic medical records (gestacional age; birth weight; anthropometry at birth, first week and week 36 post menstrual age; nutricional management; administration of probiotics), and the presence of atopic diseases at school age was corroborated by telephone interviews.

The descriptive date were summarized using medians and interquartile intervals for the continuous variables and distribution frequencies for the categorial variables. Univariate comparisons were made by the Mann-Whitney test for the continuous variables and by the chi-square test for the categorical variables. The association of comorbidities in VLBW newborns and supplementation with one type or another of probiotic was evaluated with a multinomial regression analysis, ajustando por las variables que mostraron diferencias en el análisis de homogeneidad de los grupos de estudio. The analysis was performed using IBM SPSS 20.0 for Windows software

ELIGIBILITY:
Inclusion Criteria:

* Newborn with a gestational age < or = 32 weeks and/or birth weight < or = 1500 grams.

Exclusion Criteria:

* Incomplete health history record o lack of data.
* Severe congenital anomalies.

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn with a gestational age < or = 32 weeks and/or birth weight < or = 1500 grams born at our hospital (Hospital Universitario Clínico San Cecilio, Granada) between January 2009 and December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Change incidence of atopic dermatitis in children receiving probiotics | From birth to January 2023
  The investigators will assess the presence of atopic dermatitis (itching and chronic or recurrent eczematous lesions with typical morphology and distribution) in the telephone interview.
To assess whether the combined use of breast milk and probiotics has a beneficial effect on the prevention of atopic dermatitis in children. | From birth to January 2023
  The investigators will ask patients for both attopic dermatitis involvement and a history of probiotic and breast milk administration in the neonatal period.
Identify probiotic strains that may decrease the incidence of atopic dermatitis. | From birth to January 2023
  In the group of patients who received probiotics we found two groups, one group received Lacticaseibacillus rhamnosus ATCC 53103 and the other group received the combination of Lactobacillus acidophilus ATCC 4356 + Bifidobacterium bifidum ATCC 15696. An attempt will be made to identify if there are differences between them.
Influence of caloric intake on the development of atopic dermatitis | From birth to January 2023
  The researchers will look at the medical history for caloric and macronutrient intake during the first weeks of life and assess whether it is related to differences in the development of atopic dermatitis.

CONTACTS AND LOCATIONS:
Overall Officials: José Uberos-Fernández, Mr, Principal Investigator — Hospital Clinico Universitario San Cecilio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Altobelli E, Angeletti PM, Verrotti A, Petrocelli R. The Impact of Human Milk on Necrotizing Enterocolitis: A Systematic Review and Meta-Analysis. Nutrients. 2020 May 6;12(5):1322. doi: 10.3390/nu12051322. PMID 32384652
- [Background] Bjorkander S, Carvalho-Queiroz C, Hallberg J, Persson JO, Johansson MA, Nussbaum B, Jenmalm MC, Nilsson C, Sverremark-Ekstrom E. Childhood allergy is preceded by an absence of gut lactobacilli species and higher levels of atopy-related plasma chemokines. Clin Exp Immunol. 2020 Dec;202(3):288-299. doi: 10.1111/cei.13494. Epub 2020 Aug 5. PMID 32652542
- [Background] Campos-Martinez AM, Exposito-Herrera J, Gonzalez-Bolivar M, Fernandez-Marin E, Uberos J. Evaluation of Risk and Preventive Factors for Necrotizing Enterocolitis in Premature Newborns. A Systematic Review of the Literature. Front Pediatr. 2022 May 17;10:874976. doi: 10.3389/fped.2022.874976. eCollection 2022. PMID 35656377
- [Background] Cukrowska B, Ceregra A, Maciorkowska E, Surowska B, Zegadlo-Mylik MA, Konopka E, Trojanowska I, Zakrzewska M, Bierla JB, Zakrzewski M, Kanarek E, Motyl I. The Effectiveness of Probiotic Lactobacillus rhamnosus and Lactobacillus casei Strains in Children with Atopic Dermatitis and Cow's Milk Protein Allergy: A Multicenter, Randomized, Double Blind, Placebo Controlled Study. Nutrients. 2021 Apr 1;13(4):1169. doi: 10.3390/nu13041169. PMID 33916192
- [Background] Cuna A, Morowitz MJ, Ahmed I, Umar S, Sampath V. Dynamics of the preterm gut microbiome in health and disease. Am J Physiol Gastrointest Liver Physiol. 2021 Apr 1;320(4):G411-G419. doi: 10.1152/ajpgi.00399.2020. Epub 2021 Jan 13. PMID 33439103
- [Background] Damm JA, Smith B, Greisen G, Krogfelt KA, Clausen ML, Agner T. The influence of probiotics for preterm neonates on the incidence of atopic dermatitis-results from a historically controlled cohort study. Arch Dermatol Res. 2017 May;309(4):259-264. doi: 10.1007/s00403-017-1725-4. Epub 2017 Mar 7. PMID 28271213
- [Background] David TJ, Ewing CI. Atopic eczema and preterm birth. Arch Dis Child. 1988 Apr;63(4):435-6. doi: 10.1136/adc.63.4.435. PMID 3365015
- [Background] Fanfaret IS, Boda D, Ion LM, Hosseyni D, Leru P, Ali S, Corcea S, Bumbacea R. Probiotics and prebiotics in atopic dermatitis: Pros and cons (Review). Exp Ther Med. 2021 Dec;22(6):1376. doi: 10.3892/etm.2021.10811. Epub 2021 Sep 28. PMID 34650624
- [Background] Fenton TR, Kim JH. A systematic review and meta-analysis to revise the Fenton growth chart for preterm infants. BMC Pediatr. 2013 Apr 20;13:59. doi: 10.1186/1471-2431-13-59. PMID 23601190
- [Background] Fijan S, Kolc N, Hrasovec M, Jamtvedt G, Pogacar MS, Micetic Turk D, Maver U. Single-Strain Probiotic Lactobacilli for the Treatment of Atopic Dermatitis in Children: A Systematic Review and Meta-Analysis. Pharmaceutics. 2023 Apr 17;15(4):1256. doi: 10.3390/pharmaceutics15041256. PMID 37111741
- [Background] Fuleihan RL. The hygiene hypothesis and atopic disease. Curr Opin Pediatr. 2002 Dec;14(6):676-7. doi: 10.1097/00008480-200212000-00004. No abstract available. PMID 12436033
- [Background] Gdalevich M, Mimouni D, David M, Mimouni M. Breast-feeding and the onset of atopic dermatitis in childhood: a systematic review and meta-analysis of prospective studies. J Am Acad Dermatol. 2001 Oct;45(4):520-7. doi: 10.1067/mjd.2001.114741. PMID 11568741
- [Background] Hahn WH, Kim J, Song S, Park S, Kang NM. The human milk oligosaccharides are not affected by pasteurization and freeze-drying. J Matern Fetal Neonatal Med. 2019 Mar;32(6):985-991. doi: 10.1080/14767058.2017.1397122. Epub 2017 Nov 6. PMID 29108433
- [Background] Kalliomaki M, Salminen S, Arvilommi H, Kero P, Koskinen P, Isolauri E. Probiotics in primary prevention of atopic disease: a randomised placebo-controlled trial. Lancet. 2001 Apr 7;357(9262):1076-9. doi: 10.1016/S0140-6736(00)04259-8. PMID 11297958
- [Background] Levine TA, Grunau RE, McAuliffe FM, Pinnamaneni R, Foran A, Alderdice FA. Early childhood neurodevelopment after intrauterine growth restriction: a systematic review. Pediatrics. 2015 Jan;135(1):126-41. doi: 10.1542/peds.2014-1143. PMID 25548332
- [Background] Lima PA, Carvalho Md, Costa AC, Moreira ME. Variables associated with extra uterine growth restriction in very low birth weight infants. J Pediatr (Rio J). 2014 Jan-Feb;90(1):22-7. doi: 10.1016/j.jped.2013.05.007. Epub 2013 Oct 22. PMID 24156833
- [Background] Martinez FD, Guerra S. Early Origins of Asthma. Role of Microbial Dysbiosis and Metabolic Dysfunction. Am J Respir Crit Care Med. 2018 Mar 1;197(5):573-579. doi: 10.1164/rccm.201706-1091PP. No abstract available. PMID 29048927
- [Background] Nagasaki T, Tabuchi T, Matsumoto H, Horimukai K. Age-specific associations of early daycare, older siblings, severe airway infection, and preterm birth with subsequent atopic diseases. Pediatr Allergy Immunol. 2022 Apr;33(4):e13771. doi: 10.1111/pai.13771. PMID 35470939
- [Background] Narbona Lopez E, Uberos Fernandez J, Armada Maresca MI, Couce Pico ML, Rodriguez Martinez G, Saenz de Pipaon M. [Nutrition and Metabolism Group of the Spanish Neonatology Society: recommendations and evidence for dietary supplementation with probiotics in very low birth weight infants]. An Pediatr (Barc). 2014 Dec;81(6):397.e1-8. doi: 10.1016/j.anpedi.2014.06.020. Epub 2014 Aug 6. Spanish. PMID 25106928
- [Background] Niele N, van Zwol A, Westerbeek EA, Lafeber HN, van Elburg RM. Effect of non-human neutral and acidic oligosaccharides on allergic and infectious diseases in preterm infants. Eur J Pediatr. 2013 Mar;172(3):317-23. doi: 10.1007/s00431-012-1886-2. Epub 2012 Nov 7. PMID 23132642
- [Background] Nolan LS, Rimer JM, Good M. The Role of Human Milk Oligosaccharides and Probiotics on the Neonatal Microbiome and Risk of Necrotizing Enterocolitis: A Narrative Review. Nutrients. 2020 Oct 6;12(10):3052. doi: 10.3390/nu12103052. PMID 33036184
- [Background] Nutten S. Atopic dermatitis: global epidemiology and risk factors. Ann Nutr Metab. 2015;66 Suppl 1:8-16. doi: 10.1159/000370220. Epub 2015 Apr 24. PMID 25925336
- [Background] Olesen AB, Ellingsen AR, Olesen H, Juul S, Thestrup-Pedersen K. Atopic dermatitis and birth factors: historical follow up by record linkage. BMJ. 1997 Apr 5;314(7086):1003-8. doi: 10.1136/bmj.314.7086.1003. PMID 9112844
- [Background] Olsen R, Greisen G, Schroder M, Brok J. Prophylactic Probiotics for Preterm Infants: A Systematic Review and Meta-Analysis of Observational Studies. Neonatology. 2016;109(2):105-12. doi: 10.1159/000441274. Epub 2015 Dec 2. PMID 26624488
- [Background] Panduru M, Salavastru CM, Panduru NM, Tiplica GS. Birth weight and atopic dermatitis: systematic review and meta-analyis. Acta Dermatovenerol Croat. 2014;22(2):91-6. PMID 25102793
- [Background] Pincus M, Keil T, Rucke M, Bruenahl C, Magdorf K, Klapp BF, Douglas AJ, Paus R, Wahn U, Arck P. Fetal origin of atopic dermatitis. J Allergy Clin Immunol. 2010 Jan;125(1):273-5.e1-4. doi: 10.1016/j.jaci.2009.10.057. No abstract available. PMID 20109756
- [Background] Plummer EL, Chebar Lozinsky A, Tobin JM, Uebergang JB, Axelrad C, Garland SM, Jacobs SE, Tang MLK; ProPrems Study Group. Postnatal probiotics and allergic disease in very preterm infants: Sub-study to the ProPrems randomized trial. Allergy. 2020 Jan;75(1):127-136. doi: 10.1111/all.14088. Epub 2019 Nov 8. PMID 31608448
- [Background] Rudzki E, Samochocki Z, Rebandel P, Saciuk E, Galecki W, Raczka A, Szmurlo A. Frequency and significance of the major and minor features of Hanifin and Rajka among patients with atopic dermatitis. Dermatology. 1994;189(1):41-6. doi: 10.1159/000246781. PMID 8003784
- [Background] Rzehak P, Wijga AH, Keil T, Eller E, Bindslev-Jensen C, Smit HA, Weyler J, Dom S, Sunyer J, Mendez M, Torrent M, Vall O, Bauer CP, Berdel D, Schaaf B, Chen CM, Bergstrom A, Fantini MP, Mommers M, Wahn U, Lau S, Heinrich J; GA(2)LEN-WP 1.5 Birth Cohorts. Body mass index trajectory classes and incident asthma in childhood: results from 8 European Birth Cohorts--a Global Allergy and Asthma European Network initiative. J Allergy Clin Immunol. 2013 Jun;131(6):1528-36. doi: 10.1016/j.jaci.2013.01.001. Epub 2013 Feb 10. PMID 23403049
- [Background] Samuels N, van de Graaf R, Been JV, de Jonge RC, Hanff LM, Wijnen RM, Kornelisse RF, Reiss IK, Vermeulen MJ. Necrotising enterocolitis and mortality in preterm infants after introduction of probiotics: a quasi-experimental study. Sci Rep. 2016 Aug 22;6:31643. doi: 10.1038/srep31643. PMID 27545195
- [Background] Sherman PM, Cabana M, Gibson GR, Koletzko BV, Neu J, Veereman-Wauters G, Ziegler EE, Walker WA. Potential roles and clinical utility of prebiotics in newborns, infants, and children: proceedings from a global prebiotic summit meeting, New York City, June 27-28, 2008. J Pediatr. 2009 Nov;155(5):S61-70. doi: 10.1016/j.jpeds.2009.08.022. PMID 19840609
- [Background] Simpson A, Brough HA, Haider S, Belgrave D, Murray CS, Custovic A. Early-life inhalant allergen exposure, filaggrin genotype, and the development of sensitization from infancy to adolescence. J Allergy Clin Immunol. 2020 Mar;145(3):993-1001. doi: 10.1016/j.jaci.2019.08.041. Epub 2019 Oct 17. PMID 31629803
- [Background] Steffensen FH, Sorensen HT, Gillman MW, Rothman KJ, Sabroe S, Fischer P, Olsen J. Low birth weight and preterm delivery as risk factors for asthma and atopic dermatitis in young adult males. Epidemiology. 2000 Mar;11(2):185-8. doi: 10.1097/00001648-200003000-00018. PMID 11021618
- [Background] Thureen PJ. Early aggressive nutrition in very preterm infants. Nestle Nutr Workshop Ser Pediatr Program. 2007;59:193-204; discussion 204-8. doi: 10.1159/000098536. PMID 17245100
- [Background] Trikamjee T, Comberiati P, D'Auria E, Peroni D, Zuccotti GV. Nutritional Factors in the Prevention of Atopic Dermatitis in Children. Front Pediatr. 2021 Jan 12;8:577413. doi: 10.3389/fped.2020.577413. eCollection 2020. PMID 33585361
- [Background] Uberos J. Perinatal microbiota: review of its importance in newborn health. Arch Argent Pediatr. 2020 Jun;118(3):e265-e270. doi: 10.5546/aap.2020.eng.e265. English, Spanish. PMID 32470263
- [Background] Uberos J, Aguilera-Rodriguez E, Jerez-Calero A, Molina-Oya M, Molina-Carballo A, Narbona-Lopez E. Probiotics to prevent necrotising enterocolitis and nosocomial infection in very low birth weight preterm infants. Br J Nutr. 2017 Apr;117(7):994-1000. doi: 10.1017/S0007114517000769. Epub 2017 Apr 26. PMID 28443531
- [Background] Uberos J, Campos-Martinez A, Fernandez-Marin E, Millan IC, Lopez AR, Blanca-Jover E. Effectiveness of two probiotics in preventing necrotising enterocolitis in a cohort of very-low-birth-weight premature new-borns. Benef Microbes. 2022 Feb 28;13(1):25-31. doi: 10.3920/BM2021.0088. Epub 2021 Nov 18. PMID 34794372
- [Background] Voigt J, Lele M. Lactobacillus rhamnosus Used in the Perinatal Period for the Prevention of Atopic Dermatitis in Infants: A Systematic Review and Meta-Analysis of Randomized Trials. Am J Clin Dermatol. 2022 Nov;23(6):801-811. doi: 10.1007/s40257-022-00723-x. Epub 2022 Sep 26. PMID 36161401
- [Background] Yang YW, Tsai CL, Lu CY. Exclusive breastfeeding and incident atopic dermatitis in childhood: a systematic review and meta-analysis of prospective cohort studies. Br J Dermatol. 2009 Aug;161(2):373-83. doi: 10.1111/j.1365-2133.2009.09049.x. Epub 2009 Feb 23. PMID 19239469
- [Background] Zachariassen G. Nutrition, growth, and allergic diseases among very preterm infants after hospital discharge. Dan Med J. 2013 Feb;60(2):B4588. PMID 23461996
- See also: Uberos, J., Narbona, E., Gormaz, M., Lines, M., Rodríguez, G., Saenz de Pipaón, M. and Couce, M., 2017b. Nutrición parenteral en el recién nacido prematuro de muy bajo peso. Propuesta de un protocolo de actuación tras revisión de la evidencia científica. — https://www.seneo.es/images/site/publicaciones/libros/Nutricion_parenteral.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT06035835/Prot_SAP_000.pdf